CLINICAL TRIAL: NCT06474741
Title: Both Sides Now: Using Computer Vision and App-based Intervention for Prediction and Prevention of Infant Torticollis and Plagiocephaly
Brief Title: Using Technology for Prediction and Prevention of Infant Torticollis and Plagiocephaly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Staten Island, the City University of New York (Other)
Collaborators: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CStatenIslandCUNY
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Torticollis
Keywords: prevention
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): in-app twice-weekly parent notification about torticollis and head turn asymmetries
  Interventions: Behavioral: in-app notification
- control (No Intervention): in-app twice-weekly parent notification about general infant development

INTERVENTIONS:
Behavioral: in-app notification — Parents will receive bi-weekly prompts in a baby monitor app to change infant's orientation within crib, allow for tummy time several times per day, alternate the side from which infants are fed, alternate the side the infant faces during carrying, and in general note any side preferences of the infant so that positioning can assist in symmetry.
  Arms: intervention

SUMMARY:
The goal of this clinical trial is to test whether an app-based intervention can reduce the likelihood of a torticollis diagnosis in infants. The main question[s] it aims to answer are:

* whether an app can successfully deliver an intervention to parents of young infants
* whether parents who learn about torticollis will increase behaviors intended to prevent torticollis compared to parents who learn about general infant development

Participants will complete a monthly survey for 6 months asking about their parenting behaviors. Researchers will compare parents who receive notifications about torticollis with parents who receive notifications about general infant development to see if increased knowledge of torticollis leads to preventive behavior.

ELIGIBILITY:
Inclusion Criteria:

* any parent with an infant under a month old who can answer a survey in English

Exclusion Criteria:

* infant already has a diagnosis of torticollis or plagiocephaly

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
symmetry score | baseline and 4 months
  extent of infant's head turn asymmetry

SECONDARY OUTCOMES:
gaze asymmetry score | 6 months
  extent of infant's eye gaze asymmetry
time spent in focused attention | 6 months
# of bouts of focused attention | 6 months
correlation between computer vision algorithm & manual coding for infants' head turns | 4 months
Correlate computer vision score with clinical test of symmetry | 4 months

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie results reported in published articles, after deidentification, as well as the study protocol, statistical analysis plan, and informed consent form, will be available beginning 9 months and ending 5 years following publication.
  Only investigators whose proposed use of the data has been approved by a learned intermediary shall have access to conduct analyses as approved in the proposal.